CLINICAL TRIAL: NCT02770729
Title: Use of Intracameral Moxifloxacin for the Prevention of Acute Endophthalmitis Following Cataract Surgery: a Controlled and Randomized Clinical Trial
Brief Title: Evaluation of Efficacy and Safety of Intracameral Moxifloxacin for Prevention of Postcataract Endophthalmitis.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Mathias Violante Mélega, MD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Moxi-Unicamp
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Endophthalmitis
Keywords: intracameral moxifloxacin; endophthalmitis; Vigamox; endothelial cell density
MeSH Terms: conditions — Endophthalmitis | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intracameral moxifloxacin (Active Comparator): Intracameral injection of 0.5% moxifloxacin at conclusion of cataract surgery (150 micrograms)
  Interventions: Drug: Moxifloxacin
- No injection of moxifloxacin (Sham Comparator): No injection of moxifloxacin at conclusion of cataract surgery
  Interventions: Drug: No injection of moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — Intracameral injection of moxifloxacin at conclusion of cataract surgery
  Other Names: Vigamox
  Arms: Intracameral moxifloxacin
Drug: No injection of moxifloxacin — No intracameral injection of moxifloxacin at conclusion of cataract surgery
  Other Names: No Injection
  Arms: No injection of moxifloxacin

SUMMARY:
There has thus far been only one randomized and masked clinical trial in the world to evaluate the efficacy of the intraoperative intracameral injection of antibiotics with the objective of preventing endophthalmitis following cataract surgery. The ESCRS study from 2007 confirmed that the intracameral use of cefuroxime reduced the incidence of endophthalmitis approximately fivefold. Unlike in Europe, where this drug came to be widely used after the 2007 results, cefuroxime is not commercially available in Brazil. Many studies around the world have substituted cefuroxime with moxifloxacin, which is a drug that is easily found around the world in eye drop form. It is widely used in postoperative regimens in cases of ophthalmologic surgeries, and it is free of preservatives that are toxic to intraocular structures (corneal endothelial cells). Three studies (all respective) found that the intracameral use of moxifloxacin is safe and effective for preventing endophthalmitis following cataract surgery; however, no controlled, randomized, and masked clinical trials have been performed with this objective. If this trial confirms its hypothesis (a reduction in the incidence of endophthalmitis following cataract surgery) and if minimal side effects are reported, moxifloxacin may be an option for routine intracameral use during cataract surgery, thus reducing cases of endophthalmitis and consequent cases of blindness.

DETAILED DESCRIPTION:
Patients who are diagnosed with cataracts and for whom surgery is indicated shall be evaluated in terms of their visual acuity and refractive error and via biomicroscopy, automated keratometry (Auto Kerato Refractometer KR 8000® Alcon), Goldmann applanation tonometry, fundoscopy, biometric assessment (Ocuscan RxP® Alcon or Lenstar LS900® Haag-Streit International), and specular microscopy of the cornea (EM-3000® Tomey) to count the corneal endothelial cells. Each cataract case shall be classified based on the Lens Opacities Classification System III (LOCS III).

Patients who choose to sign the informed consent form after being informed of all of the aspects of the surgery and this trial shall be randomly divided into 2 groups that shall be approximately equal in size and stratified by gender. Group A shall receive an intracameral injection of 0.03ml of 0.5% moxifloxacin (150 micrograms in 0.03 ml) at the end of the cataract surgery, followed by the use of a 0.5% moxifloxacin in eye drop form associated with 0.1% dexamethasone before the bandage is applied. Group B shall not receive the intracameral moxifloxacin injection at the end of the cataract surgery; these patients shall receive only 0.5% moxifloxacin in eye drop form associated with 0.1% dexamethasone before the bandage is applied.

The cataract surgery shall be performed using the standards followed by the Department of Ophthalmology at São Paulo State University, Campinas (UNICAMP). It shall be performed by second-, third-, and fourth-year ophthalmology residents and by attendings when cases are more complex. Preoperative pupil dilation shall be performed through the use of 10% phenylephrine and 1% tropicamide 3 times in five-minute increments. The anesthesiology technique used shall depend on each case and shall be either topical anesthesia, peribulbar anesthesia, sub-Tenon anesthesia, or general anesthesia. Skin sterilization shall be performed using an aqueous solution of 10% povidone-iodine. After the sterile surgical field is established and the eyelashes are isolated, 4 eye drops containing 5% povidone-iodine shall be administered in the conjunctival sac with subsequent irrigation using a 10% balanced salt solution. In cases of allergy to povidone-iodine, an aqueous solution of 0.05% chlorhexidine shall be used. The principal incision (using a clear corneal incision or the near clear approach) shall be 2.2mm to 3.0mm in length. The phacoemulsification technique shall be either the stop and chop, the phaco chop, the pre-slice, the pre-chop, or the divide and conquer; it shall be applied through the use of the Infiniti® or the Laureate® phacoemulsifier (Alcon), with an AcrySof® intraocular foldable lens (Alcon). In cases of posterior capsule rupture and vitreous loss, a complication that increases the chance of endophthalmitis,3,4,15 a mechanical or manual anterior vitrectomy shall be performed (the choice shall depend on the case). In cases of thermal burn of the principal incision or other situations in which surgical injury is not self-sealing and in which there is a consequent leak of the aqueous humor and an inability to keep the anterior chamber in adequate dimensions, the incision shall be sutured using Mononylon 10.0.

The moxifloxacin injection shall be prepared by a trained nurse or physician: 0.03ml (150 micrograms) of 0.5% moxifloxacin as an ophthalmic solution (Vigamox®) shall be aspirated. The eye drop bottles shall be opened at the moment of preparation with a 0.3ml coupled syringe (Terumo®) through the use of an asseptic technique. The solution shall then be injected into the anterior chamber via paracentesis as the last step in the phacoemulsification surgery. The patients from the two groups shall receive 0.5% moxifloxacin drops associated with 0.1% dexamethasone after the surgery is completed and before the bandage is applied. The postoperative prescription shall consist of 0.5% moxifloxacin associated with 0.1% dexamethasone. Administration shall begin 3 hours after the surgery is completed and should continue every 3 hours for 7 days (except when the patient is sleeping). After the 7th postoperative day, 0.1% dexamethasone without association with moxifloxacin shall be prescribed. Its application shall be gradually reduced over the course of 3 weeks according to each individual's inflammatory response.

Patients from both groups shall be masked, while the surgeons and ophthalmologists who perform the postoperative examinations will not. In suspected cases of endophthalmitis, an independent ophthalmologist from a retina and vitreous practice shall perform the patient's examination without knowing whether the patient belongs to Group A or Group B. This independent ophthalmologist shall then recommend the most adequate course of action. Endophthalmitis treatment shall follow the usual protocol. The postoperative consults shall be held on the 1st, 7th, 30th, and 45th postoperative days and shall include evaluations of visual acuity (7th, 30th, and 45th postoperative day), refractive error (30th postoperative day), biomicroscopy (1st, 7th, 30th, and 45th postoperative day), applanation tonometry (7th, 30th, and 45th postoperative day), keratometry (30th postoperative day), fundoscopy (30th, and 45th post operative day), and endothelial cell counts (45th postoperative day).

The diagnosis of acute endophthalmitis following cataract surgery shall initially be clinical and shall be considered presumed until the microorganism in question can be identified through laboratory exams.

Cases of sudden worsening in vision after cataract surgery (up to 6 weeks post-operation) and associated with pain, palpebral edema, red eye, corneal edema, signs of intraocular inflammation (such as inflammatory cells in the vitreous, anterior chamber reaction, hypopyon, and effects on the vitreous detected via ultrasound) shall be considered suspected cases of endophthalmitis. These patients shall undergo aqueous humor and vitreous humor sample collections under surgical conditions in order to detect the etiological agent (bacterioscopy and culture). In addition, broad-spectrum empiric antibiotic therapy shall be employed due to the high morbidity of this complication.

The diagnosis of endophthalmitis shall be based on the laboratory confirmation of the presence of microorganisms in aqueous humor or vitreous humor samples, or by the evaluation of the clinical findings (presumed endophthalmitis) if an etiological agent is not identified in a case that is characteristic of endophthalmitis.

Based on the 0.3% frequency of endophthalmitis in 2015 in cataract surgeries without prophylactic treatment with antibiotics at the Clinical Hospital of São Paulo State University, Campinas (UNICAMP), a one-tailed confidence interval of 95%, 80% power, an exposed :non-exposed correlation of 1:1, and a null endophthalmitis frequency were applied to the group treated with the antibiotic. Approximately 2,600 volunteers will be needed for each group.

The trial shall be suspended with a difference between the two groups that is inferior to a type I error (α) of 4% is found in a pre-analysis with 25%, 50%, 62.5%, 75%, and 87.5%of the total number of patients to be analyzed.

Scheduled surgeries shall be distributed in blocks of four volunteers stratified by gender. This step will ensure that each block of four patients will include two volunteers from each group.

After the attribution of the interventions, each patient shall be masked to the type of intervention. The surgeons and the ophthalmologists who will perform the postoperative examinations (usually the surgeons themselves) will not be masked. In suspected cases of endophthalmitis, an independent ophthalmologist from a retina and vitreous practice shall evaluate the patient and recommend the most adequate course of action.

Measures of central tendency and dispersion shall be determined using averages and standard deviations. Tests shall be performed to detect differences between the categorical variables. The chi-square test and Fisher's exact test shall be used. One-way ANOVA and Student's t-test shall be used to detect differences between quantitative variables. The results of these analyses shall be considered significant if the p-value is lower than 5%. The statistical analysis shall be performed within the EpiInfoTM 2000 software (Centers for Disease Control and Prevention, Atlanta, Georgia, USA) and within SPSS®,

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of visually significant cataract

Exclusion Criteria

* Moxifloxacin allergy
* Traumatic cataract with ocular perforation
* Cataract surgery associated with other procedures, such as glaucoma filtering surgery, vitreoretinal surgery, and cornea surgery
* Signs of ocular or periocular infection
* Advanced glaucoma
* Severe dry eye

Ages: 40 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3640 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Endophthalmitis incidence | 45 days
  Endophthalmitis incidence in each group

SECONDARY OUTCOMES:
Endothelial cell count | 45 days
  Endothelial cell count loss in each group

CONTACTS AND LOCATIONS:
Overall Officials: Mathias V Mélega, MD, Principal Investigator — University of Campinas
Locations (1):
- Mathias Violante Mélega, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arieta CE, de Oliveira DF, Lupinacci AP, Novaes P, Paccola M, Jose NK, Limburg H. Cataract remains an important cause of blindness in Campinas, Brazil. Ophthalmic Epidemiol. 2009 Jan-Feb;16(1):58-63. doi: 10.1080/09286580802575032. PMID 19191183
- [Background] Melo GB, Bispo PJ, Regatieri CV, Yu MC, Pignatari AC, Hofling-Lima AL. Incidence of endophthalmitis after cataract surgery (2002-2008) at a Brazilian university-hospital. Arq Bras Oftalmol. 2010 Nov-Dec;73(6):505-7. doi: 10.1590/s0004-27492010000600007. PMID 21271024
- [Background] Friling E, Lundstrom M, Stenevi U, Montan P. Six-year incidence of endophthalmitis after cataract surgery: Swedish national study. J Cataract Refract Surg. 2013 Jan;39(1):15-21. doi: 10.1016/j.jcrs.2012.10.037. PMID 23245359
- [Background] Endophthalmitis Study Group, European Society of Cataract & Refractive Surgeons. Prophylaxis of postoperative endophthalmitis following cataract surgery: results of the ESCRS multicenter study and identification of risk factors. J Cataract Refract Surg. 2007 Jun;33(6):978-88. doi: 10.1016/j.jcrs.2007.02.032. PMID 17531690
- [Background] Kowalski RP, Romanowski EG, Mah FS, Yates KA, Gordon YJ. Intracameral Vigamox (moxifloxacin 0.5%) is non-toxic and effective in preventing endophthalmitis in a rabbit model. Am J Ophthalmol. 2005 Sep;140(3):497-504. doi: 10.1016/j.ajo.2005.04.015. PMID 16083841
- [Background] Kim SY, Park YH, Lee YC. Comparison of the effect of intracameral moxifloxacin, levofloxacin and cefazolin on rabbit corneal endothelial cells. Clin Exp Ophthalmol. 2008 May;36(4):367-70. doi: 10.1111/j.1442-9071.2008.01771.x. PMID 18700925
- [Background] Lane SS, Osher RH, Masket S, Belani S. Evaluation of the safety of prophylactic intracameral moxifloxacin in cataract surgery. J Cataract Refract Surg. 2008 Sep;34(9):1451-9. doi: 10.1016/j.jcrs.2008.05.034. PMID 18721703
- [Background] Espiritu CR, Caparas VL, Bolinao JG. Safety of prophylactic intracameral moxifloxacin 0.5% ophthalmic solution in cataract surgery patients. J Cataract Refract Surg. 2007 Jan;33(1):63-8. doi: 10.1016/j.jcrs.2006.09.019. PMID 17189795
- [Background] Matsuura K, Miyoshi T, Suto C, Akura J, Inoue Y. Efficacy and safety of prophylactic intracameral moxifloxacin injection in Japan. J Cataract Refract Surg. 2013 Nov;39(11):1702-6. doi: 10.1016/j.jcrs.2013.05.036. Epub 2013 Sep 18. PMID 24054967
- [Background] Matsuura K, Suto C, Akura J, Inoue Y. Comparison between intracameral moxifloxacin administration methods by assessing intraocular concentrations and drug kinetics. Graefes Arch Clin Exp Ophthalmol. 2013 Aug;251(8):1955-9. doi: 10.1007/s00417-013-2294-7. Epub 2013 Apr 2. PMID 23546399
- [Background] Javitt JC. Intracameral Antibiotics Reduce the Risk of Endophthalmitis after Cataract Surgery: Does the Preponderance of the Evidence Mandate a Global Change in Practice? Ophthalmology. 2016 Feb;123(2):226-231. doi: 10.1016/j.ophtha.2015.12.011. No abstract available. PMID 26802702
- [Background] Shorstein NH, Winthrop KL, Herrinton LJ. Decreased postoperative endophthalmitis rate after institution of intracameral antibiotics in a Northern California eye department. J Cataract Refract Surg. 2013 Jan;39(1):8-14. doi: 10.1016/j.jcrs.2012.07.031. Epub 2012 Oct 2. PMID 23036356
- [Background] Haripriya A, Chang DF, Namburar S, Smita A, Ravindran RD. Efficacy of Intracameral Moxifloxacin Endophthalmitis Prophylaxis at Aravind Eye Hospital. Ophthalmology. 2016 Feb;123(2):302-308. doi: 10.1016/j.ophtha.2015.09.037. Epub 2015 Oct 30. PMID 26522705